CLINICAL TRIAL: NCT00005123
Title: Honolulu Heart Program
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 902
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2004-09

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Cerebrovascular Accident; Heart Diseases; Heart Failure, Congestive; Myocardial Infarction; Asthma; Emphysema; Lung Diseases, Obstructive; Aortic Aneurysm, Abdominal; Bronchitis; Dementia; Hypertension; Chronic Obstructive Pulmonary Disease; Heart Failure
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Stroke; Heart Diseases; Heart Failure; Myocardial Infarction; Asthma; Emphysema; Lung Diseases, Obstructive; Aortic Aneurysm, Abdominal; Bronchitis; Dementia; Hypertension; Pulmonary Disease, Chronic Obstructive

SUMMARY:
To investigate coronary heart disease and stroke among American men of Japanese ancestry who were living on the island of Oahu in 1965. Morbidity and mortality surveillance of the original cohort is continuing.

DETAILED DESCRIPTION:
BACKGROUND:

The Honolulu Heart Program was initiated to verify reports that men of Japanese ancestry living in the United States had a much higher risk of coronary heart disease and a lower risk of stroke than Japanese men in Japan. The Honolulu Heart Program was actually a component of the larger NI-HON-SAN Study. The NI-HON-SAN Study (from the acronyms Nippon, Honolulu, and San Francisco) was initiated in 1965. The populations under investigation included members of the Honolulu Heart Program as well as men of Japanese ancestry born between 1900 and 1919 and residing in Japan and San Francisco.

In the Honolulu Heart Program, 11,148 men were identified of whom 8,006 participated in baseline examinations between 1965 and 1968. The 1965 - 1968 examination included a detailed medical and social history with specific inquiries about smoking, alcohol consumption, diet, and physical activity. A physical examination focussed on the cardiovascular system; laboratory tests included hematocrit, serum cholesterol, triglyceride, uric acid, glucose determination, and urinalysis. A twelve lead electrocardiogram and lung function testing revealed that 301 men had evidence of coronary heart disease and 111 had a stroke. The prevalence of coronary heart disease was slightly higher than in the comparable population in Japan, but the incidence rate during the first two-year period of follow-up was twice as high in Honolulu as in Japan. Stroke prevalence was much higher in Japan than in the Honolulu cohort, with a threefold difference. The Honolulu Japanese men were more obese, ate a more Westernized diet with a higher amount of animal protein, saturated fat, and sucrose and a smaller amount of complex carbohydrates. They had higher levels of serum cholesterol, triglyceride, uric acid, and glucose than Japanese men in Japan. Cigarette smoking was more common in the Japanese cohort, while the proportion of heavy smokers was greater in the Honolulu cohort. Alcohol consumption in the Japanese cohort was twice that of the Honolulu cohort. There were no differences in mean blood pressure or prevalence of hypertension. Repeat examinations were performed near the second and sixth anniversaries of the initial examinations. The six year follow-up data identified 294 new cases of coronary heart disease and 133 new cases of stroke. Between 1970 and 1972 some 2,800 of the cohort were examined and had lipoprotein determinations performed as part of the NHLBI Lipoprotein Phenotyping Project. Survivors of the lipoprotein cohort were reexamined between 1975 and 1978 near the tenth anniversary of their initial examination and again between 1980 and 1982.

In 1985, the program was enlarged to make a comparative analysis of the 12-year incidence of coronary heart disease in the Japanese and Hawaii study cohort of the original NI-HON-SAN Study, to sample 400 offspring of the study cohort ages 45 to 60 years and to complete nutrient indicators for association with blood pressure in a manner consistent with the United States-Japan study of nutrition and blood pressure. Resulting data were compared with a comparable selected group of Japanese men and with the parents of the offspring to examine familial associations. Pulmonary function data were recorded and analyzed for association with other risk factors, respiratory disease, and other major chronic diseases.

Beginning in March 1993 and continuing through December 1994, the National Institute on Aging, with its own funds, investigated aging and dementia among Honolulu Heart Program participants.

Beginning in March 1997, the study was supported by U01HL56274.

DESIGN NARRATIVE:

In this prospective cohort study, the hospital discharge rosters of all general hospitals on the Island of Oahu were reviewed twice yearly as part of the morbidity and mortality surveillance. The appropriate chart materials were abstracted for review by study physicians for evidence of myocardial infarction and stroke. Beginning in 1986, both old and new hospital discharge records were reviewed for the additional endpoints of congestive heart failure, aortic aneurysm, bronchitis, emphysema, asthma, chronic obstructive lung disease, dementia, organic brain syndrome, and Parkinson's disease. Deaths were monitored by following obituary columns as well as reviewing death certificates from the State Health Department. There was daily contact with hospitals to find out about impending autopsies in which study personnel could participate. However, only 20-25 percent of the deaths had protocol autopsies.

The fifth and final complete examination of the surviving cohort concluded in Spring, 1996 under a contract with the National Institute on Aging. While the emphasis of this exam was the investigation of dementia, NHLBI funded the recording of blood pressures and ECGs as well as the continued surveillance for morbidity and mortality. A cooperative agreement extends the surveillance for an additional five years. As part of the close-out phase of the study, frozen blood samples collected since the study's inception have been sent to a repository in Rockville, MD. A review board for screening prospective users of this resource holds quarterly meetings.

As the study group includes both migrants from Japan and Hawaii-born men, there is a spectrum of cultural lifestyles and varying grades of acculturation which are being examined as risk factors for cardiovascular and other chronic diseases. The existing baseline and follow-up examination data and the surveillance information on the incidence of most major diseases provide opportunities for a great variety of research projects concerning the predictors of cardiovascular disease, as well as studies of the broader concepts of health and disease in the aging population. The low out-migration rate and the well-defined sources of medical care have provided an ideal setting for maintaining disease morbidity and mortality surveillance; nearly 100 per cent of hospital discharge episodes have been recorded. As the study participants range in age from 75-95 in 1996, the rates of coronary heart disease, stroke, and other chronic diseases are increasing rapidly and thus are providing a large number of disease endpoints for study. Other Institutes are also currently supporting activities which utilize the original cohort.

Stored sera provide an opportunity to test new ideas and etiologic hypotheses using both prospective and case-control study designs. Protocol autopsy information can now be utilized to examine relationships among risk factors, clinical manifestations of CHD, and stroke and pathological evidence of atherosclerosis.

Beginning in 1997, a cooperative agreement extends the surveillance for an additional five years through February, 2002. As part of the close-out of the study, frozen blood samples collected since the study's inception have been sent to a repository in Rockville, Maryland.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1965-07; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Overall Officials: J. Curb — Kuakini Medical Center; Jess Curb — Kuakini Medical Center

REFERENCES:
- [Background] Rhoads GG. Hemoglobin A1c reproducibility. Ann Intern Med. 1980 Apr;92(4):574. doi: 10.7326/0003-4819-92-4-574. No abstract available. PMID 7362177
- [Background] McGee D, Rhoads G, Feinleib M: The Logistic Function. A Model for Assessing Risk of Heart Disease. In Proceedings of the Fourteenth Hawaii International Conference on System Sciences. Edited by B. Shriver et al. Honolulu, Hawaii, University of Hawaii Press pp 722-740, 1981
- [Background] Blackwelder WC, Kagan A, Gordon T, Rhoads GG. Comparison of methods for diagnosing angina pectoris: the Honolulu heart study. Int J Epidemiol. 1981 Sep;10(3):211-5. doi: 10.1093/ije/10.3.211. PMID 7287281
- [Background] Gordon T, Kagan A, Garcia-Palmieri M, Kannel WB, Zukel WJ, Tillotson J, Sorlie P, Hjortland M. Diet and its relation to coronary heart disease and death in three populations. Circulation. 1981 Mar;63(3):500-15. doi: 10.1161/01.cir.63.3.500. PMID 7460234
- [Background] Kagan A, McGee DL, Yano K, Rhoads GG, Nomura A. Serum cholesterol and mortality in a Japanese-American population: the Honolulu Heart program. Am J Epidemiol. 1981 Jul;114(1):11-20. doi: 10.1093/oxfordjournals.aje.a113157. PMID 7246518
- [Background] Kagan A, Yano K, Rhoads GG, McGee DL. Alcohol and cardiovascular disease: the Hawaiian experience. Circulation. 1981 Sep;64(3 Pt 2):III 27-31. PMID 7261298
- [Background] Reed D, McGee D, Yano K. Biological and social correlates of blood pressure among Japanese men in Hawaii. Hypertension. 1982 May-Jun;4(3):406-14. doi: 10.1161/01.hyp.4.3.406. PMID 7068196
- [Background] Yano K, Kagan A, McGee D, Rhoads GG. Glucose intolerance and nine-year mortality in Japanese men in Hawaii. Am J Med. 1982 Jan;72(1):71-80. doi: 10.1016/0002-9343(82)90580-0. PMID 7058826
- [Background] McGee D, Rhoads G, Hankin J, Yano K, Tillotson J. Within-person variability of nutrient intake in a group of Hawaiian men of Japanese ancestry. Am J Clin Nutr. 1982 Oct;36(4):657-63. doi: 10.1093/ajcn/36.4.657. PMID 7124667
- [Background] Reed D, McGee D, Cohen J, Yano K, Syme SL, Feinleib M. Acculturation and coronary heart disease among Japanese men in Hawaii. Am J Epidemiol. 1982 Jun;115(6):894-905. doi: 10.1093/oxfordjournals.aje.a113377. PMID 7091147
- [Background] Kagan A, Yano K, McGee D, Rhoads GG: Epidemiology of Glucose Intolerance in Hawaii Japanese Men. Excerpta Medica. In: Genetic-Enviornmental Interaction in Diabetes Mellitus, Proceedings of the Third Symposium on Diabetes Mellitus in Asia and Oceania; Honolulu Feb 6-7, 1981; ISBN Elsevier North Holland, (International Congress Series No. 549, pp 51-56, 1982
- [Background] Hulley SB, Rhoads GG. The plasma lipoproteins as risk factors: comparison of electrophoretic and ultracentrifugation results. Metabolism. 1982 Aug;31(8):773-7. doi: 10.1016/0026-0495(82)90074-9. PMID 6954343
- [Background] Yamamoto L, Yano K, Rhoads GG. Characteristics of joggers among Japanese men in Hawaii. Am J Public Health. 1983 Feb;73(2):147-52. doi: 10.2105/ajph.73.2.147. PMID 6849472
- [Background] Yano K, McGee D, Reed DM. The impact of elevated blood pressure upon 10-year mortality among Japanese men in Hawaii: the Honolulu Heart Program. J Chronic Dis. 1983;36(8):569-79. doi: 10.1016/0021-9681(83)90145-5. PMID 6885958
- [Background] Reed D, McGee D, Yano K. Trends of coronary heart disease among men of Japanese ancestry in Hawaii. J Community Health. 1983 Spring;8(3):149-59. doi: 10.1007/BF01666450. PMID 6875040
- [Background] Carter C, McGee D, Reed D, Yano K, Stemmermann G. Hematocrit and the risk of coronary heart disease: the Honolulu Heart Program. Am Heart J. 1983 Apr;105(4):674-9. doi: 10.1016/0002-8703(83)90493-3. No abstract available. PMID 6837420
- [Background] Reed D, McGee D, Yano K, Feinleib M. Social networks and coronary heart disease among Japanese men in Hawaii. Am J Epidemiol. 1983 Apr;117(4):384-96. doi: 10.1093/oxfordjournals.aje.a113557. PMID 6837553
- [Background] Rhoads GG, Feinleib M. Serum triglyceride and risk of coronary heart disease, stroke, and total mortality in Japanese-American men. Arteriosclerosis. 1983 Jul-Aug;3(4):316-22. doi: 10.1161/01.atv.3.4.316. PMID 6882286
- [Background] Rhoads GG, Kagan A. The relation of coronary disease, stroke, and mortality to weight in youth and in middle age. Lancet. 1983 Mar 5;1(8323):492-5. doi: 10.1016/s0140-6736(83)92189-x. PMID 6131209
- [Background] Rao DC, Williams WR, McGue M, Morton NE, Gulbrandsen CL, Rhoads GG, Kagan A, Laskarzewski P, Glueck CJ, Russell JM. Cultural and biological inheritance of plasma lipids. Am J Phys Anthropol. 1983 Sep;62(1):33-49. doi: 10.1002/ajpa.1330620107. PMID 6624899
- [Background] Williams WR, Morton NE, Rao DC, Gulbrandsen CL, Rhoads GG, Kagan A. Family resemblance for fasting blood glucose in a population of Japanese Americans. Clin Genet. 1983 Apr;23(4):287-93. doi: 10.1111/j.1399-0004.1983.tb01878.x. PMID 6851219
- [Background] Reed DM, Feinleib M. Changing patterns of cardiovascular disease in the Pacific Basin: report of an international workshop. J Community Health. 1983 Spring;8(3):182-205. doi: 10.1007/BF01666453. No abstract available. PMID 6875043
- [Background] Reed D: Social Stress, Social Support and Hypertension Among Japanese Men in Hawaii. In Proceedings of the Second Intercontinental Symposium on Hypertension and the Japanese. Molokai, Hawaii. Japan, Medical Tribune, pp 21-30, 1983
- [Background] Reed D, McGee D, Yano K. Psychosocial processes and general susceptibility to chronic disease. Am J Epidemiol. 1984 Mar;119(3):356-70. doi: 10.1093/oxfordjournals.aje.a113754. PMID 6702812
- [Background] Yano K, Reed DM, McGee DL. Ten-year incidence of coronary heart disease in the Honolulu Heart Program. Relationship to biologic and lifestyle characteristics. Am J Epidemiol. 1984 May;119(5):653-66. doi: 10.1093/oxfordjournals.aje.a113787. PMID 6720665
- [Background] Stemmermann GN, Hayashi T, Resch JA, Chung CS, Reed DM, Rhoads GG. Risk factors related to ischemic and hemorrhagic cerebrovascular disease at autopsy: the Honolulu Heart Study. Stroke. 1984 Jan-Feb;15(1):23-8. doi: 10.1161/01.str.15.1.23. PMID 6695427
- [Background] Carter C, McGee D, Yano K. Morbidity and mortality rates in Okinawan Japanese vs. mainland Japanese: the Honolulu Heart Program. Hum Biol. 1984 May;56(2):339-53. No abstract available. PMID 6489984
- [Background] Stemmermann GN, Heilbrun L, Nomura A, Rhoads GG, Glober GA. Late mortality after partial gastrectomy. Int J Epidemiol. 1984 Sep;13(3):299-303. doi: 10.1093/ije/13.3.299. PMID 6490300
- [Background] McGee DL, Reed DM, Yano K, Kagan A, Tillotson J. Ten-year incidence of coronary heart disease in the Honolulu Heart Program. Relationship to nutrient intake. Am J Epidemiol. 1984 May;119(5):667-76. doi: 10.1093/oxfordjournals.aje.a113788. PMID 6720666
- [Background] Takeya Y, Popper JS, Shimizu Y, Kato H, Rhoads GG, Kagan A. Epidemiologic studies of coronary heart disease and stroke in Japanese men living in Japan, Hawaii and California: incidence of stroke in Japan and Hawaii. Stroke. 1984 Jan-Feb;15(1):15-23. doi: 10.1161/01.str.15.1.15. PMID 6695420
- [Background] McGee D, Reed D, Yano K. The results of logistic analyses when the variables are highly correlated: an empirical example using diet and CHD incidence. J Chronic Dis. 1984;37(9-10):713-9. doi: 10.1016/0021-9681(84)90040-7. PMID 6501543
- [Background] McGee D, Reed D, Stemmerman G, Rhoads G, Yano K, Feinleib M. The relationship of dietary fat and cholesterol to mortality in 10 years: the Honolulu Heart Program. Int J Epidemiol. 1985 Mar;14(1):97-105. doi: 10.1093/ije/14.1.97. PMID 3988448
- [Background] Joffres M, Reed DM, Nomura AM. Psychosocial processes and cancer incidence among Japanese men in Hawaii. Am J Epidemiol. 1985 Apr;121(4):488-500. doi: 10.1093/oxfordjournals.aje.a114027. PMID 4014140
- [Background] Reed D, McGee D, Yano K, Hankin J. Diet, blood pressure, and multicollinearity. Hypertension. 1985 May-Jun;7(3 Pt 1):405-10. PMID 3838968
- [Background] Benfante R, Reed D, Brody J. Biological and social predictors of health in an aging cohort. J Chronic Dis. 1985;38(5):385-95. doi: 10.1016/0021-9681(85)90134-1. PMID 3998053
- [Background] Kagan A, Popper JS, Rhoads GG, Yano K. Dietary and other risk factors for stroke in Hawaiian Japanese men. Stroke. 1985 May-Jun;16(3):390-6. doi: 10.1161/01.str.16.3.390. PMID 4002255
- [Background] Reed D, Benfante R. Predictors of health in men of Japanese ancestry in Hawaii. Hawaii Med J. 1985 Aug;44(8):307-8. No abstract available. PMID 4055359
- [Background] Yano K, Reed DM, Kagan A. Coronary heart disease, hypertension and stroke among Japanese-American men in Hawaii: the Honolulu Heart Program. Hawaii Med J. 1985 Aug;44(8):297-300, 312. No abstract available. PMID 4055357
- [Background] Cohen JB, Reed D. The type A behavior pattern and coronary heart disease among Japanese men in Hawaii. J Behav Med. 1985 Dec;8(4):343-52. doi: 10.1007/BF00848368. PMID 4093972
- [Background] Curb JD, Reed DM, Kautz JA, Yano K. Coffee, caffeine, and serum cholesterol in Japanese men in Hawaii. Am J Epidemiol. 1986 Apr;123(4):648-55. doi: 10.1093/oxfordjournals.aje.a114284. PMID 3953543
- [Background] Donahue RP, Abbott RD, Reed DM, Yano K. Alcohol and hemorrhagic stroke. The Honolulu Heart Program. JAMA. 1986 May 2;255(17):2311-4. PMID 3959320
- [Background] Reed D, Yano K, Kagan A. Lipids and lipoproteins as predictors of coronary heart disease, stroke, and cancer in the Honolulu Heart Program. Am J Med. 1986 May;80(5):871-8. doi: 10.1016/0002-9343(86)90631-5. PMID 3706375
- [Background] Yano K, Reed DM, Curb JD, Hankin JH, Albers JJ. Biological and dietary correlates of plasma lipids and lipoproteins among elderly Japanese men in Hawaii. Arteriosclerosis. 1986 Jul-Aug;6(4):422-33. doi: 10.1161/01.atv.6.4.422. PMID 3488054
- [Background] Abbott RD, Yin Y, Reed DM, Yano K. Risk of stroke in male cigarette smokers. N Engl J Med. 1986 Sep 18;315(12):717-20. doi: 10.1056/NEJM198609183151201. PMID 3748080
- [Background] Curb JD, Reed DM, Yano K, Kautz JA, Albers JJ. Plasma lipids and lipoproteins in elderly Japanese-American men. J Am Geriatr Soc. 1986 Nov;34(11):773-80. doi: 10.1111/j.1532-5415.1986.tb03980.x. PMID 3771975
- [Background] Rhoads GG, Dahlen G, Berg K, Morton NE, Dannenberg AL. Lp(a) lipoprotein as a risk factor for myocardial infarction. JAMA. 1986 Nov 14;256(18):2540-4. PMID 2945939
- [Background] Abbott RD, Donahue RP, MacMahon SW, Reed DM, Yano K. Diabetes and the risk of stroke. The Honolulu Heart Program. JAMA. 1987 Feb 20;257(7):949-52. PMID 3806877
- [Background] Reed D, Labarthe D, Chen KM, Stallones R. A cohort study of amyotrophic lateral sclerosis and parkinsonism-dementia on Guam and Rota. Am J Epidemiol. 1987 Jan;125(1):92-100. doi: 10.1093/oxfordjournals.aje.a114515. PMID 3788958
- [Background] Donahue RP, Abbott RD, Bloom E, Reed DM, Yano K. Central obesity and coronary heart disease in men. Lancet. 1987 Apr 11;1(8537):821-4. doi: 10.1016/s0140-6736(87)91605-9. PMID 2882231
- [Background] Joffres MR, Reed DM, Yano K. Relationship of magnesium intake and other dietary factors to blood pressure: the Honolulu heart study. Am J Clin Nutr. 1987 Feb;45(2):469-75. doi: 10.1093/ajcn/45.2.469. PMID 3812346
- [Background] Reed DM, MacLean CJ, Hayashi T. Predictors of atherosclerosis in the Honolulu Heart Program. I. Biologic, dietary, and lifestyle characteristics. Am J Epidemiol. 1987 Aug;126(2):214-25. doi: 10.1093/aje/126.2.214. PMID 3605050
- [Background] MacLean CJ, Reed DM. Predictors of atherosclerosis in the Honolulu Heart Program. II. Adjustment for autopsy bias. Am J Epidemiol. 1987 Aug;126(2):226-36. doi: 10.1093/aje/126.2.226. PMID 3605051
- [Background] Coffee consumption and the incidence of coronary heart disease. N Engl J Med. 1987 Apr 9;316(15):945-7. doi: 10.1056/NEJM198704093161513. No abstract available. PMID 3821843
- [Background] Donahue RP, Abbott RD, Reed DM, Yano K. Postchallenge glucose concentration and coronary heart disease in men of Japanese ancestry. Honolulu Heart Program. Diabetes. 1987 Jun;36(6):689-92. doi: 10.2337/diab.36.6.689. PMID 3569669
- [Background] Reed D, Yano K. Epidemiological studies of hypertension among elderly Japanese and Japanese Americans. Asia Pac J Public Health. 1987;1(2):49-56. doi: 10.1177/101053958700100210. No abstract available. PMID 3452393
- [Background] Reed DM: Predictors of a Long Healthy Life Among Japanese Men in Hawaii. In: Prevention of Cardiovascular Diseases: an Approach to Active Long Life. Yamori Y, Lenfant C (Eds). Elsevier Science Publishers, pp 225-234, 1987
- [Background] Yano K, McCarthy LJ, Reed DM, Kagan A. Postmortem findings in sudden and non-sudden deaths among Japanese-American men in Hawaii. Am J Med. 1987 Dec;83(6):1037-44. doi: 10.1016/0002-9343(87)90939-9. PMID 3503573
- [Background] Yano K, MacLean CJ, Reed DM, Shimizu Y, Sasaki H, Kodama K, Kato H, Kagan A. A comparison of the 12-year mortality and predictive factors of coronary heart disease among Japanese men in Japan and Hawaii. Am J Epidemiol. 1988 Mar;127(3):476-87. doi: 10.1093/oxfordjournals.aje.a114824. PMID 3341354
- [Background] Donahue RP, Abbott RD, Reed DM, Yano K. Physical activity and coronary heart disease in middle-aged and elderly men: the Honolulu Heart Program. Am J Public Health. 1988 Jun;78(6):683-5. doi: 10.2105/ajph.78.6.683. PMID 3369600
- [Background] Marcus EB, Buist AS, Curb JD, MacLean CJ, Reed DM, Johnson LR, Yano K. Correlates of FEV1 and prevalence of pulmonary conditions in Japanese-American men. Am Rev Respir Dis. 1988 Dec;138(6):1398-404. doi: 10.1164/ajrccm/138.6.1398. PMID 3202494
- [Background] Marcus EB, MacLean CJ, Curb JD, Johnson LR, Vollmer WM, Buist AS. Reference values for FEV1 in Japanese-American men from 45 to 68 years of age. Am Rev Respir Dis. 1988 Dec;138(6):1393-7. doi: 10.1164/ajrccm/138.6.1393. PMID 3202493
- [Background] Miller FD, Reed DM, MacLean CJ. A prospective study of mortality and morbidity among carpenters in the Honolulu Heart Program Cohort. J Occup Med. 1988 Nov;30(11):879-82. doi: 10.1097/00043764-198811000-00015. PMID 3230436
- [Background] Reed DM, Resch JA, Hayashi T, MacLean C, Yano K. A prospective study of cerebral artery atherosclerosis. Stroke. 1988 Jul;19(7):820-5. doi: 10.1161/01.str.19.7.820. PMID 3388454
- [Background] Reed DM, Strong JP, Hayashi T, Newman WP 3rd, Tracy RE, Guzman MA, Stemmermann GN. Comparison of two measures of atherosclerosis in a prospective epidemiology study. Arteriosclerosis. 1988 Nov-Dec;8(6):782-7. doi: 10.1161/01.atv.8.6.782. PMID 3196221
- [Background] Knutsen R, Knutsen SF, Curb JD, Reed DM, Kautz JA, Yano K. Predictive value of resting electrocardiograms for 12-year incidence of stroke in the Honolulu Heart Program. Stroke. 1988 May;19(5):555-9. doi: 10.1161/01.str.19.5.555. PMID 3363587
- [Background] Trombold JC, Moellering RC Jr, Kagan A. Epidemiological aspects of coronary heart disease and cerebrovascular disease: the Honolulu Heart Program. Hawaii Med J. 1966 Jan-Feb;25(3):231-4. No abstract available. PMID 5906867
- [Background] Worth RM, Kagan A. Ascertainment of men of Japanese ancestry in Hawaii through World War II Selective Service registration. J Chronic Dis. 1970 Nov;23(5):389-97. doi: 10.1016/0021-9681(70)90022-6. No abstract available. PMID 5492969
- [Background] Kagan A, Rhoads GG, Zeegen PD, Nichaman MZ. Coronary heart disease among men of Japanese ancestry in Hawaii. The Honolulu Heart study. Isr J Med Sci. 1971 Dec;7(12):1573-7. No abstract available. PMID 5144601
- [Background] Belsky JL, Kagan A, Syme SL: Epidemiologic Studies of Coronary Heart Disease and Stroke in Japanese Men Living in Japan, Hawaii and California: Research Plan. ABCC TR 12-71, 1971
- [Background] Sano T, Yokoyama M, Rhoads GG. Clinical significance of 1 -antitrypsin level--a preliminary evaluation among Japanese men. Hawaii Med J. 1972 Jan-Feb;31(1):27-32. No abstract available. PMID 5015359
- [Background] Gould SE, Hayashi T, Tashiro T, Tanimura A, Nakashima T, Shohoji T. Coronary heart disease and stroke. Atherosclerosis in Japanese men in Hiroshima, Japan and Honolulu, Hawaii. Arch Pathol. 1972 Feb;93(2):98-102. No abstract available. PMID 5009022
- [Background] Rhoads GG, Zeegen PD, Glober GA, Boelling GM: The Epidemiology of Pterygium a High Risk Population. Transactions of Pacific Coast Oto-Ophthalmological Society pp 163-173, 1972
- [Background] Tillotson JL, Kato H, Nichaman MZ, Miller DC, Gay ML, Johnson KG, Rhoads GG. Epidemiology of coronary heart disease and stroke in Japanese men living in Japan, Hawaii, and California: methodology for comparison of diet. Am J Clin Nutr. 1973 Feb;26(2):177-84. doi: 10.1093/ajcn/26.2.177. No abstract available. PMID 4703052
- [Background] Kato H, Tillotson J, Nichaman MZ, Rhoads GG, Hamilton HB. Epidemiologic studies of coronary heart disease and stroke in Japanese men living in Japan, Hawaii and California. Am J Epidemiol. 1973 Jun;97(6):372-85. doi: 10.1093/oxfordjournals.aje.a121518. No abstract available. PMID 4713933
- [Background] Kagan A: The World Wide Investigation of the Epidemiology of Coronary Heart Disease. J Hiroshima Med Assoc 26:10:1145-1157, 1973
- [Background] Glober GA, Rhoads GG, Liu F, Kagan A. Long term results of gastrectomy with respect to blood lipids, blood pressure, weight and living habits. Ann Surg. 1974 Jun;179(6):896-901. doi: 10.1097/00000658-197406000-00013. PMID 4835509
- [Background] Phillips RL, Lilienfeld AM, Diamond EL, Kagan A. Frequency of coronary heart disease and cerebrovascular accidents in parents and sons of coronary heart disease index cases and controls. Am J Epidemiol. 1974 Aug;100(2):87-100. doi: 10.1093/oxfordjournals.aje.a112021. No abstract available. PMID 4852095
- [Background] Gordon T, Garcia-Palmieri MR, Kagan A, Kannel WB, Schiffman J. Differences in coronary heart disease in Framingham, Honolulu and Puerto Rico. J Chronic Dis. 1974 Sep;27(7-8):329-44. doi: 10.1016/0021-9681(74)90013-7. No abstract available. PMID 4436425
- [Background] Kagan A, Harris BR, Winkelstein W Jr, Johnson KG, Kato H, Syme SL, Rhoads GG, Gay ML, Nichaman MZ, Hamilton HB, Tillotson J. Epidemiologic studies of coronary heart disease and stroke in Japanese men living in Japan, Hawaii and California: demographic, physical, dietary and biochemical characteristics. J Chronic Dis. 1974 Sep;27(7-8):345-64. doi: 10.1016/0021-9681(74)90014-9. No abstract available. PMID 4436426
- [Background] Gordon T, Kagan A, Rhoads G. Letters to the editor: Relative weights in different populations. Am J Clin Nutr. 1975 Apr;28(4):304-5. doi: 10.1093/ajcn/28.4.304. No abstract available. PMID 1119426
- [Background] Yano K, Peskoe SM, Rhoads GG, Moore JO, Kagan A. Left axis deviation and left anterior hemiblock among 8,000 Japanese-American men. Am J Cardiol. 1975 Jun;35(6):809-15. doi: 10.1016/0002-9149(75)90116-2. PMID 1130290
- [Background] Syme SL, Marmot MG, Kagan A, Kato H, Rhoads G. Epidemiologic studies of coronary heart disease and stroke in Japanese men living in Japan, Hawaii and California: introduction. Am J Epidemiol. 1975 Dec;102(6):477-80. doi: 10.1093/oxfordjournals.aje.a112185. PMID 1202949
- [Background] Worth RM, Kato H, Rhoads GG, Kagan K, Syme SL. Epidemiologic studies of coronary heart disease and stroke in Japanese men living in Japan, Hawaii and California: mortality. Am J Epidemiol. 1975 Dec;102(6):481-90. doi: 10.1093/oxfordjournals.aje.a112186. PMID 1202950
- [Background] Nichaman MZ, Hamilton HB, Kagan A, Grier T, Sacks T, Syme SL. Epidemiologic studies of coronary heart disease and stroke in Japanese men living in Japan, Hawaii and California: distribution of biochemical risk factors. Am J Epidemiol. 1975 Dec;102(6):491-501. doi: 10.1093/oxfordjournals.aje.a112187. PMID 1202951
- [Background] Winkelstein W Jr, Kagan A, Kato H, Sacks ST. Epidemiologic studies of coronary heart disease and stroke in Japanese men living in Japan, Hawaii and California: blood pressure distributions. Am J Epidemiol. 1975 Dec;102(6):502-13. doi: 10.1093/oxfordjournals.aje.a112188. PMID 1202952
- [Background] Marmot MG, Syme SL, Kagan A, Kato H, Cohen JB, Belsky J. Epidemiologic studies of coronary heart disease and stroke in Japanese men living in Japan, Hawaii and California: prevalence of coronary and hypertensive heart disease and associated risk factors. Am J Epidemiol. 1975 Dec;102(6):514-25. doi: 10.1093/oxfordjournals.aje.a112189. PMID 1202953
- [Background] Rhoads GG, Kagan A, Yano K. Usefulness of community surveillance for the ascertainment of coronary heart disease and stroke. Int J Epidemiol. 1975 Dec;4(4):265-70. doi: 10.1093/ije/4.4.265. PMID 23682412
- [Background] Kagan A, Gordon T, Rhoads GG, Schiffman JC. Some factors related to coronary heart disease incidence in Honolulu Japanese men: the Honolulu Heart Study. Int J Epidemiol. 1975 Dec;4(4):271-9. doi: 10.1093/ije/4.4.271. PMID 23682413
- [Background] Hankin JH, Nomura A, Rhoads GG. Dietary patterns among men of Japanese ancestry in Hawaii. Cancer Res. 1975 Nov;35(11 Pt. 2):3259-64. PMID 1192401
- [Background] Winkelstein W Jr: Cooperative Studies of Blood Pressure in Japanese in Japan, Hawaii and the United States. In Epidemiology and Control of Hypertension Paul O (Ed.) Miami: Symposia Specialists, pp 101-114, 1975
- [Background] Rhoads GG, Gulbrandsen CL, Kagan A. Serum lipoproteins and coronary heart disease in a population study of Hawaii Japanese men. N Engl J Med. 1976 Feb 5;294(6):293-8. doi: 10.1056/NEJM197602052940601. PMID 173994
- [Background] Kagan A: Epidemiology of Hypertension and Stroke in Oceania. In Hypertension and Stroke Control in the Community Hatano S, Shigematsu I, Strasser T (Eds.) Geneva: World Health Organization, pp 97-105, 1976
- [Background] Stemmermann GN, Steer A, Rhoads GG, Lee K, Hayashi T, Nakashima T, Keehn R. A comparative pathology study of myocardial lesions and atherosclerosis in Japanese men living in Hiroshima, Japan and Honolulu, Hawaii. Lab Invest. 1976 Jun;34(6):592-600. PMID 132567
- [Background] Kagan A, Popper J, Rhoads GG, Takeya Y, Kato H, Brown-Goode G, Marmot MG: Epidemiologic Studies of Coronary Heart Disease and Stroke in Japanese Men Living in Japan, Hawaii, and California: Prevalence of Stroke. In Cerebrovascular Diseases, Tenth Princeton Conference Scheinberg P (Ed.) New York: Raven Press, pp 267-277, 1976
- [Background] Robertson TL, Kato H, Rhoads GG, Kagan A, Marmot M, Syme SL, Gordon T, Worth RM, Belsky JL, Dock DS, Miyanishi M, Kawamoto S. Epidemiologic studies of coronary heart disease and stroke in Japanese men living in Japan, Hawaii and California. Incidence of myocardial infarction and death from coronary heart disease. Am J Cardiol. 1977 Feb;39(2):239-43. doi: 10.1016/s0002-9149(77)80197-5. PMID 835482
- [Background] Robertson TL, Kato H, Gordon T, Kagan A, Rhoads GG, Land CE, Worth RM, Belsky JL, Dock DS, Miyanishi M, Kawamoto S. Epidemiologic studies of coronary heart disease and stroke in Japanese men living in Japan, Hawaii and California. Coronary heart disease risk factors in Japan and Hawaii. Am J Cardiol. 1977 Feb;39(2):244-9. doi: 10.1016/s0002-9149(77)80198-7. PMID 835483
- [Background] Rhoads GG, Klein K, Yano K, Preston H. The earlobe crease--sign of obesity in middle-aged Japanese men. Hawaii Med J. 1977 Mar;36(3):74-7. No abstract available. PMID 845018
- [Background] Morton NE, MacLean CJ, Kagan A, Gulbrandsen CL, Rhoads GG, Yee S, Lew R. Commingling in distributions of lipids and related variables. Am J Hum Genet. 1977 Jan;29(1):52-9. PMID 835575
- [Background] Yano K, Rhoads G, Kagan A. Epidemiology of serum uric acid among 8000 Japanese-American men in Hawaii. J Chronic Dis. 1977 Mar;30(3):171-84. doi: 10.1016/0021-9681(77)90083-2. No abstract available. PMID 849973
- [Background] Castelli WP, Cooper GR, Doyle JT, Garcia-Palmieri M, Gordon T, Hames C, Hulley SB, Kagan A, Kuchmak M, McGee D, Vicic WJ. Distribution of triglyceride and total, LDL and HDL cholesterol in several populations: a cooperative lipoprotein phenotyping study. J Chronic Dis. 1977 Mar;30(3):147-69. doi: 10.1016/0021-9681(77)90082-0. No abstract available. PMID 191465
- [Background] Castelli WP, Doyle JT, Gordon T, Hames CG, Hjortland MC, Hulley SB, Kagan A, Zukel WJ. HDL cholesterol and other lipids in coronary heart disease. The cooperative lipoprotein phenotyping study. Circulation. 1977 May;55(5):767-72. doi: 10.1161/01.cir.55.5.767. PMID 191215
- [Background] Castelli WP, Doyle JT, Gordon T, Hames CG, Hjortland MC, Hulley SB, Kagan A, Zukel WJ. Alcohol and blood lipids. The cooperative lipoprotein phenotyping study. Lancet. 1977 Jul 23;2(8030):153-5. doi: 10.1016/s0140-6736(77)90176-3. PMID 69778
- [Background] Yano K, Rhoads GG, Kagan A. Coffee, alcohol and risk of coronary heart disease among Japanese men living in Hawaii. N Engl J Med. 1977 Aug 25;297(8):405-9. doi: 10.1056/NEJM197708252970801. PMID 882109
- [Background] Takeya Y, Kato H, Kagan A, Popper J, Rhoads GG, Browne Goode G, Marmot M: Epidemiologic Study of Stroke in Japanese Men Living in Japan, Hawaii and California: Prevalence of Stroke. In Gene-Environment Interaction in Common Diseases Inouye E, Nishimura H (Eds.) University of Tokyo Press, pp 15-18, 1977
- [Background] Roberts A, Kagan A, Rhoads GG, Pierce JA, Bruce RM. Antitrypsin and chronic obstructive pulmonary disease among Japanese-American men. Chest. 1977 Oct;72(4):489-91. doi: 10.1378/chest.72.4.489. PMID 302780
- [Background] Gulbrandsen CL, Morton NE, Rhoads GG, Kagan A, Lew R. Behavioral, social, and physiological determinants of lipoprotein concentrations. Soc Biol. 1977 Winter;24(4):289-93. doi: 10.1080/19485565.1977.9988299. No abstract available. PMID 607401
- [Background] Yano K, Rhoads GG, Kagan A, Tillotson J. Dietary intake and the risk of coronary heart disease in Japanese men living in Hawaii. Am J Clin Nutr. 1978 Jul;31(7):1270-9. doi: 10.1093/ajcn/31.7.1270. PMID 665576
- [Background] Rhoads GG, Blackwelder WC, Stemmermann GN, Hayashi T, Kagan A. Coronary risk factors and autopsy findings in Japanese-American men. Lab Invest. 1978 Mar;38(3):304-11. PMID 633854
- [Background] Morton NE, Gulbrandsen CL, Rhoads GG, Kagan A. The Lp lipoprotein in Japanese. Clin Genet. 1978 Oct;14(4):207-12. doi: 10.1111/j.1399-0004.1978.tb02132.x. PMID 699359
- [Background] Rhoads GG, Morton NE, Gulbrandsen CL, Kagan A. Sinking pre-beta lipoprotein and coronary heart disease in Japanese-American men in Hawaii. Am J Epidemiol. 1978 Nov;108(5):350-6. doi: 10.1093/oxfordjournals.aje.a112631. PMID 215032
- [Background] Morton NE, Gulbrandsen CL, Rhoads GG, Kagan A, Lew R. Major loci for lipoprotein concentrations. Am J Hum Genet. 1978 Nov;30(6):583-9. PMID 747186
- [Background] Gulbrandsen CL, Morton NE, Rao DC, Rhoads GG, Kagan A. Determinants of plasma uric acid. Hum Genet. 1979 Sep;50(3):307-12. doi: 10.1007/BF00399397. PMID 489016
- [Background] Yano K, Blackwelder WC, Kagan A, Rhoads GG, Cohen JB, Marmot MG. Childhood cultural experience and the incidence of coronary heart disease in Hawaii Japanese men. Am J Epidemiol. 1979 Apr;109(4):440-50. doi: 10.1093/oxfordjournals.aje.a112702. PMID 443242
- [Background] Kagan A, Yano K, Rhoads GG, Kato H. Is the reported high mortality from cerebrovascular disease in Japan really an artefact? J Chronic Dis. 1979;32(1-2):153-6. doi: 10.1016/0021-9681(79)90043-2. No abstract available. PMID 447775
- [Background] Mitsuyama Y, Thompson LR, Hayashi T, Lee KK, Keehn RJ, Resch JA, Steer A. Autopsy study of cerebrovascular disease in Japanese men who lived in Hiroshima, Japan, and Honolulu, Hawaii. Stroke. 1979 Jul-Aug;10(4):389-95. doi: 10.1161/01.str.10.4.389. PMID 505476
- [Background] Steer A, Lee SS, Stemmermann GN, Yamamoto T, Rhoads GG, Lee KK. Autopsy study of small cardiac scars in Japanese men who lived in Hiroshima, Japan and Honolulu, Hawaii. Lab Invest. 1979 Dec;41(6):538-45. PMID 513645
- [Background] Cohen JB, Syme SL, Jenkins CD, Kagan A, Zyzanski SJ. Cultural context of type A behavior and risk for CHD: a study of Japanese American males. J Behav Med. 1979 Dec;2(4):375-84. doi: 10.1007/BF00844741. PMID 548580
- [Background] Rao DC, Morton NE, Gulbrandsen CL, Rhoads GG, Kagan A, Yee S. Cultural and biological determinants of lipoprotein concentrations. Ann Hum Genet. 1979 May;42(4):467-77. doi: 10.1111/j.1469-1809.1979.tb00680.x. PMID 475334
- [Background] Morton NE, Gulbrandsen CL, Rao DC, Rhoads GG, Kagan A. Determinants of blood pressure in Japanese-American Families. Hum Genet. 1980 Feb;53(2):261-6. doi: 10.1007/BF00273508. PMID 7358393
- [Background] Kagan A, Popper JS, Rhoads GG. Factors related to stroke incidence in Hawaii Japanese men. The Honolulu Heart Study. Stroke. 1980 Jan-Feb;11(1):14-21. doi: 10.1161/01.str.11.1.14. PMID 6444469
- [Background] Rhoads GG, Popper JS, Kagan A, Yano K. Incidence of transient cerebral ischemic attack in Hawaii Japanese men. The Honolulu Heart Study. Stroke. 1980 Jan-Feb;11(1):21-6. doi: 10.1161/01.str.11.1.21. PMID 7355424
- [Background] Blackwelder WC, Yano K, Rhoads GG, Kagan A, Gordon T, Palesch Y. Alcohol and mortality: the Honolulu Heart Study. Am J Med. 1980 Feb;68(2):164-9. doi: 10.1016/0002-9343(80)90350-2. PMID 7355889
- [Background] Kagan A, Marmot MG, Kato H: The Ni-Hon-San Study of Cardiovascular Disease Epidemiology: Population Characteristics and Epidemiology of Stroke. In Epidemiology of Arterial Blood Pressure. Kesteloot H, Joossens JV (Eds.). The Hague/Boston/London: Martinus Nijhoff, pp 423-436, 1980, 0000
- [Background] Marmot MG, Kagan A, Kato H: Hypertension and Heart Disease in the Ni-Hon-San Study. In Epidemiology of Arterial Blood Pressure. Kesteloot H, Joossens JV (Eds.). The Hague/Boston/London: Martinus Nijhoff, pp 437-452, 1980
- [Background] Knutsen R, Knutsen SF, Curb JD, Reed DM, Kautz JA, Yano K. The predictive value of resting electrocardiograms for 12-year incidence of coronary heart disease in the Honolulu Heart Program. J Clin Epidemiol. 1988;41(3):293-302. doi: 10.1016/0895-4356(88)90134-5. PMID 3339383
- [Background] Phillips GB, Yano K, Stemmermann GN. Serum sex hormone levels and myocardial infarction in the Honolulu Heart Program. Pitfalls in prospective studies on sex hormones. J Clin Epidemiol. 1988;41(12):1151-6. doi: 10.1016/0895-4356(88)90018-2. PMID 3210063
- [Background] Tracy RE, MacLean CJ, Reed DM, Hayashi T, Gandia M, Strong JP. Blood pressure, nephrosclerosis, and age autopsy findings from the Honolulu Heart Program. Mod Pathol. 1988 Nov;1(6):420-7. PMID 3065780
- [Background] Marcus EB, Curb JD, MacLean CJ, Reed DM, Yano K. Pulmonary function as a predictor of coronary heart disease. Am J Epidemiol. 1989 Jan;129(1):97-104. doi: 10.1093/oxfordjournals.aje.a115128. PMID 2910076
- [Background] Marcus EB, Yano K, MacLean CJ. Regression of Q waves following acute myocardial infarction. Am J Epidemiol. 1989 Jan;129(1):105-11. doi: 10.1093/oxfordjournals.aje.a115099. PMID 2910054
- [Background] Benfante RJ, Reed DM, MacLean CJ, Yano K. Risk factors in middle age that predict early and late onset of coronary heart disease. J Clin Epidemiol. 1989;42(2):95-104. doi: 10.1016/0895-4356(89)90082-6. PMID 2918328
- [Background] Kagan A, Yano K, Reed DM, MacLean CJ. Predictors of sudden cardiac death among Hawaiian-Japanese men. Am J Epidemiol. 1989 Aug;130(2):268-77. doi: 10.1093/oxfordjournals.aje.a115333. PMID 2750726
- [Background] Marcus EB, Buist AS, Maclean CJ, Yano K. Twenty-year trends in mortality from chronic obstructive pulmonary disease: the Honolulu Heart Program. Am Rev Respir Dis. 1989 Sep;140(3 Pt 2):S64-8. doi: 10.1164/ajrccm/140.3_Pt_2.S64. PMID 2782762
- [Background] Criqui MH, Langer RD, Reed DM. Dietary alcohol, calcium, and potassium. Independent and combined effects on blood pressure. Circulation. 1989 Sep;80(3):609-14. doi: 10.1161/01.cir.80.3.609. PMID 2766513
- [Background] Reed DM, LaCroix AZ, Karasek RA, Miller D, MacLean CA. Occupational strain and the incidence of coronary heart disease. Am J Epidemiol. 1989 Mar;129(3):495-502. doi: 10.1093/oxfordjournals.aje.a115160. PMID 2916542
- [Background] Benfante R, Reed D, MacLean C, Kagan A. Response bias in the Honolulu Heart Program. Am J Epidemiol. 1989 Dec;130(6):1088-100. doi: 10.1093/oxfordjournals.aje.a115436. PMID 2589302
- [Background] Benfante R, Reed D. Is elevated serum cholesterol level a risk factor for coronary heart disease in the elderly? JAMA. 1990 Jan 19;263(3):393-6. PMID 2294305
- [Background] Joffres MR, MacLean CJ, Reed DM, Yano K, Benfante R. Potential bias due to prevalent diseases in prospective studies. Int J Epidemiol. 1990 Jun;19(2):459-65. doi: 10.1093/ije/19.2.459. PMID 2376462
- [Background] Curb JD, Reed DM, Miller FD, Yano K. Health status and life style in elderly Japanese men with a long life expectancy. J Gerontol. 1990 Sep;45(5):S206-11. doi: 10.1093/geronj/45.5.s206. PMID 2394921
- [Background] Reed DM. The paradox of high risk of stroke in populations with low risk of coronary heart disease. Am J Epidemiol. 1990 Apr;131(4):579-88. doi: 10.1093/oxfordjournals.aje.a115542. PMID 2316492
- [Background] Ross GW, Abbott RD, Petrovitch H, Morens DM, Grandinetti A, Tung KH, Tanner CM, Masaki KH, Blanchette PL, Curb JD, Popper JS, White LR. Association of coffee and caffeine intake with the risk of Parkinson disease. JAMA. 2000 May 24-31;283(20):2674-9. doi: 10.1001/jama.283.20.2674. PMID 10819950
- [Background] Yano K, Grove JS, Masaki KH, White LR, Petrovitch H, Chen R, Teng EL, Ross GW, Rodriguez BL, Curb JD. The effects of childhood residence in Japan and testing language on cognitive performance in late life among Japanese American men in Hawaii. J Am Geriatr Soc. 2000 Feb;48(2):199-204. doi: 10.1111/j.1532-5415.2000.tb03912.x. PMID 10682950
- [Background] Hakim AA, Curb JD, Burchfiel CM, Rodriguez BL, Sharp DS, Yano K, Abbott RD. Screening for coronary heart disease in elderly men based on current and past cholesterol levels. J Clin Epidemiol. 1999 Dec;52(12):1257-65. doi: 10.1016/s0895-4356(99)00130-4. PMID 10580790
- [Background] Yano K, Kodama K, Shimizu Y, Chyou PH, Sharp DS, Tracy RP, Rodriguez BL, Curb JD, Kusumi S. Plasma fibrinogen and its correlates in elderly Japanese men living in Japan and Hawaii. J Clin Epidemiol. 1999 Dec;52(12):1201-6. doi: 10.1016/s0895-4356(99)00095-5. PMID 10580783
- [Background] Rodriguez BL, Lau N, Burchfiel CM, Abbott RD, Sharp DS, Yano K, Curb JD. Glucose intolerance and 23-year risk of coronary heart disease and total mortality: the Honolulu Heart Program. Diabetes Care. 1999 Aug;22(8):1262-5. doi: 10.2337/diacare.22.8.1262. PMID 10480768
- [Background] Ross GW, Petrovitch H, White LR, Masaki KH, Li CY, Curb JD, Yano K, Rodriguez BL, Foley DJ, Blanchette PL, Havlik R. Characterization of risk factors for vascular dementia: the Honolulu-Asia Aging Study. Neurology. 1999 Jul 22;53(2):337-43. doi: 10.1212/wnl.53.2.337. PMID 10430423
- [Background] Hakim AA, Curb JD, Petrovitch H, Rodriguez BL, Yano K, Ross GW, White LR, Abbott RD. Effects of walking on coronary heart disease in elderly men: the Honolulu Heart Program. Circulation. 1999 Jul 6;100(1):9-13. doi: 10.1161/01.cir.100.1.9. PMID 10393674
- [Background] Kalmijn S, Curb JD, Rodriguez BL, Yano K, Abbott RD. The association of body weight and anthropometry with mortality in elderly men: the Honolulu Heart Program. Int J Obes Relat Metab Disord. 1999 Apr;23(4):395-402. doi: 10.1038/sj.ijo.0800832. PMID 10340818
- [Background] Curb JD, Rodriguez BL, Abbott RD, Petrovitch H, Ross GW, Masaki KH, Foley D, Blanchette PL, Harris T, Chen R, White LR. Longitudinal association of vascular and Alzheimer's dementias, diabetes, and glucose tolerance. Neurology. 1999 Mar 23;52(5):971-5. doi: 10.1212/wnl.52.5.971. PMID 10102414
- [Background] Rantanen T, Guralnik JM, Foley D, Masaki K, Leveille S, Curb JD, White L. Midlife hand grip strength as a predictor of old age disability. JAMA. 1999 Feb 10;281(6):558-60. doi: 10.1001/jama.281.6.558. PMID 10022113
- [Background] Masaki KH, Schatz IJ, Burchfiel CM, Sharp DS, Chiu D, Foley D, Curb JD. Orthostatic hypotension predicts mortality in elderly men: the Honolulu Heart Program. Circulation. 1998 Nov 24;98(21):2290-5. doi: 10.1161/01.cir.98.21.2290. PMID 9826316
- [Background] Abbott RD, Yano K, Hakim AA, Burchfiel CM, Sharp DS, Rodriguez BL, Curb JD. Changes in total and high-density lipoprotein cholesterol over 10- and 20-year periods (the Honolulu Heart Program). Am J Cardiol. 1998 Jul 15;82(2):172-8. doi: 10.1016/s0002-9149(98)00310-5. PMID 9678287
- [Background] Hakim AA, Ross GW, Curb JD, Rodriguez BL, Burchfiel CM, Sharp DS, Yano K, Abbott RD. Coffee consumption in hypertensive men in older middle-age and the risk of stroke: the Honolulu Heart Program. J Clin Epidemiol. 1998 Jun;51(6):487-94. doi: 10.1016/s0895-4356(98)00023-7. PMID 9635997
- [Background] Alagiakrishnan K, Masaki K, Schatz I, Curb JD, Blanchette P. Postural hypertension in elderly men--the Honolulu Heart Program. Hawaii Med J. 2000 Feb;59(2):48-50. PMID 10800251
- [Background] Edwards KL, Burchfiel CM, Sharp DS, Curb JD, Rodriguez BL, Fujimoto WY, LaCroix AZ, Vitiello MV, Austin MA. Factors of the insulin resistance syndrome in nondiabetic and diabetic elderly Japanese-American men. Am J Epidemiol. 1998 Mar 1;147(5):441-7. doi: 10.1093/oxfordjournals.aje.a009469. PMID 9525530
- [Background] Burchfiel CM, Sharp DS, Curb JD, Rodriguez BL, Abbott RD, Arakaki R, Yano K. Hyperinsulinemia and cardiovascular disease in elderly men: the Honolulu Heart Program. Arterioscler Thromb Vasc Biol. 1998 Mar;18(3):450-7. doi: 10.1161/01.atv.18.3.450. PMID 9514414
- [Background] Burchfiel CM, Abbott RD, Curb JD, Sharp DS, Rodriguez BL, Arakaki R, Yano K. Association of insulin levels with lipids and lipoproteins in elderly Japanese-American men. Ann Epidemiol. 1998 Feb;8(2):92-8. doi: 10.1016/s1047-2797(97)00167-1. PMID 9491933
- [Background] Hakim AA, Petrovitch H, Burchfiel CM, Ross GW, Rodriguez BL, White LR, Yano K, Curb JD, Abbott RD. Effects of walking on mortality among nonsmoking retired men. N Engl J Med. 1998 Jan 8;338(2):94-9. doi: 10.1056/NEJM199801083380204. PMID 9420340
- [Background] Sharp DS, Burchfiel CM, Curb JD, Rodriguez BL, Enright PL. The synergy of low lung function and low body mass index predicting all-cause mortality among older Japanese-American men. J Am Geriatr Soc. 1997 Dec;45(12):1464-71. doi: 10.1111/j.1532-5415.1997.tb03197.x. PMID 9400556
- [Background] Abbott RD, Sharp DS, Burchfiel CM, Curb JD, Rodriguez BL, Hakim AA, Yano K. Cross-sectional and longitudinal changes in total and high-density-lipoprotein cholesterol levels over a 20-year period in elderly men: the Honolulu Heart Program. Ann Epidemiol. 1997 Aug;7(6):417-24. doi: 10.1016/s1047-2797(97)00043-4. PMID 9279451
- [Background] Burchfiel CM, Enright PL, Sharp DS, Chyou PH, Rodriguez BL, Curb JD. Factors associated with variations in pulmonary function among elderly Japanese-American men. Chest. 1997 Jul;112(1):87-97. doi: 10.1378/chest.112.1.87. PMID 9228362
- [Background] Huang B, Rodreiguez BL, Burchfiel CM, Chyou PH, Curb JD, Sharp DS. Associations of adiposity with prevalent coronary heart disease among elderly men: the Honolulu Heart Program. Int J Obes Relat Metab Disord. 1997 May;21(5):340-8. doi: 10.1038/sj.ijo.0800410. PMID 9152734
- [Background] Masaki KH, Curb JD, Chiu D, Petrovitch H, Rodriguez BL. Association of body mass index with blood pressure in elderly Japanese American men. The Honolulu Heart Program. Hypertension. 1997 Feb;29(2):673-7. doi: 10.1161/01.hyp.29.2.673. PMID 9040455
- [Background] Chyou PH, Burchfiel CM, Yano K, Sharp DS, Rodriguez BL, Curb JD, Nomura AM. Obesity, alcohol consumption, smoking, and mortality. Ann Epidemiol. 1997 May;7(4):311-7. doi: 10.1016/s1047-2797(97)00019-7. PMID 9177115
- [Background] Curb JD, Masaki K, Rodriguez BL, Abbott RD, Burchfiel CM, Chen R, Petrovitch H, Sharp D, Yano K. Peripheral artery disease and cardiovascular risk factors in the elderly. The Honolulu Heart Program. Arterioscler Thromb Vasc Biol. 1996 Dec;16(12):1495-500. doi: 10.1161/01.atv.16.12.1495. PMID 8977454
- [Background] Burchfiel CM, Curb JD, Arakaki R, Abbott RD, Sharp DS, Rodriguez BL, Yano K. Cardiovascular risk factors and hyperinsulinemia in elderly men: the Honolulu Heart Program. Ann Epidemiol. 1996 Nov;6(6):490-7. doi: 10.1016/s1047-2797(96)00103-2. PMID 8978879
- [Background] Burchfiel CM, Abbott RD, Sharp DS, Curb JD, Rodriguez BL, Yano K. Distribution and correlates of lipids and lipoproteins in elderly Japanese-American men. The Honolulu Heart Program. Arterioscler Thromb Vasc Biol. 1996 Nov;16(11):1356-64. doi: 10.1161/01.atv.16.11.1356. PMID 8911274
- [Background] Huang B, Rodriguez BL, Burchfiel CM, Chyou PH, Curb JD, Yano K. Acculturation and prevalence of diabetes among Japanese-American men in Hawaii. Am J Epidemiol. 1996 Oct 1;144(7):674-81. doi: 10.1093/oxfordjournals.aje.a008980. PMID 8823064
- [Background] Rodriguez BL, Sharp DS, Abbott RD, Burchfiel CM, Masaki K, Chyou PH, Huang B, Yano K, Curb JD. Fish intake may limit the increase in risk of coronary heart disease morbidity and mortality among heavy smokers. The Honolulu Heart Program. Circulation. 1996 Sep 1;94(5):952-6. doi: 10.1161/01.cir.94.5.952. PMID 8790031
- [Background] Rodriguez BL, Curb JD, Burchfiel CM, Huang B, Sharp DS, Lu GY, Fujimoto W, Yano K. Impaired glucose tolerance, diabetes, and cardiovascular disease risk factor profiles in the elderly. The Honolulu Heart Program. Diabetes Care. 1996 Jun;19(6):587-90. doi: 10.2337/diacare.19.6.587. PMID 8725856
- [Background] Iribarren C, Sharp DS, Curb JD, Yano K. High uric acid: a metabolic marker of coronary heart disease among alcohol abstainers. J Clin Epidemiol. 1996 Jun;49(6):673-8. doi: 10.1016/0895-4356(96)00034-0. PMID 8656229
- [Background] Burchfiel CM, Marcus EB, Sharp DS, Enright PL, Rodriguez BL, Masaki KH, Hwang LJ, Curb JD. Characteristics associated with rapid decline in forced expiratory volume. Ann Epidemiol. 1996 May;6(3):217-27. doi: 10.1016/1047-2797(96)00007-5. PMID 8827157
- [Background] Sharp DS, Curb JD, Schatz IJ, Meiselman HJ, Fisher TC, Burchfiel CM, Rodriguez BL, Yano K. Mean red cell volume as a correlate of blood pressure. Circulation. 1996 May 1;93(9):1677-84. doi: 10.1161/01.cir.93.9.1677. PMID 8653873
- [Background] Curb JD, Abbott RD, MacLean CJ, Rodriguez BL, Burchfiel CM, Sharp DS, Ross GW, Yano K. Age-related changes in stroke risk in men with hypertension and normal blood pressure. Stroke. 1996 May;27(5):819-24. doi: 10.1161/01.str.27.5.819. PMID 8623099
- [Background] Abbott RD, Curb JD, Rodriguez BL, Sharp DS, Burchfiel CM, Yano K. Effect of dietary calcium and milk consumption on risk of thromboembolic stroke in older middle-aged men. The Honolulu Heart Program. Stroke. 1996 May;27(5):813-8. doi: 10.1161/01.str.27.5.813. PMID 8623098
- [Background] Chyou PH, White LR, Yano K, Sharp DS, Burchfiel CM, Chen R, Rodriguez BL, Curb JD. Pulmonary function measures as predictors and correlates of cognitive functioning in later life. Am J Epidemiol. 1996 Apr 15;143(8):750-6. doi: 10.1093/oxfordjournals.aje.a008812. PMID 8610684
- [Background] Sharp DS, Abbott RD, Burchfiel CM, Rodriguez BL, Tracy RP, Yano K, Curb JD. Plasma fibrinogen and coronary heart disease in elderly Japanese-American men. Arterioscler Thromb Vasc Biol. 1996 Feb;16(2):262-8. doi: 10.1161/01.atv.16.2.262. PMID 8620341
- [Background] Sharp DS, Enright PL, Chiu D, Burchfiel CM, Rodriguez BL, Curb JD. Reference values for pulmonary function tests of Japanese-American men aged 71 to 90 years. Am J Respir Crit Care Med. 1996 Feb;153(2):805-11. doi: 10.1164/ajrccm.153.2.8564136.
- [Background] Curb JD, Aluli NE, Huang BJ, Sharp DS, Rodriguez BL, Burchfiel CM, Chiu D. Hypertension in elderly Japanese Americans and adult native Hawaiians. Public Health Rep. 1996;111 Suppl 2(Suppl 2):53-5. PMID 8898776
- [Background] Burchfiel CM, Curb JD, Sharp DS, Rodriguez BL, Arakaki R, Chyou PH, Yano K. Distribution and correlates of insulin in elderly men. The Honolulu Heart Program. Arterioscler Thromb Vasc Biol. 1995 Dec;15(12):2213-21. doi: 10.1161/01.atv.15.12.2213. PMID 7489245
- [Background] Burchfiel CM, Laws A, Benfante R, Goldberg RJ, Hwang LJ, Chiu D, Rodriguez BL, Curb JD, Sharp DS. Combined effects of HDL cholesterol, triglyceride, and total cholesterol concentrations on 18-year risk of atherosclerotic disease. Circulation. 1995 Sep 15;92(6):1430-6. doi: 10.1161/01.cir.92.6.1430. PMID 7664423
- [Background] Young DR, Masaki KH, Curb JD. Associations of physical activity with performance-based and self-reported physical functioning in older men: the Honolulu Heart Program. J Am Geriatr Soc. 1995 Aug;43(8):845-54. doi: 10.1111/j.1532-5415.1995.tb05525.x. PMID 7636090
- [Background] Burchfiel CM, Marcus EB, Curb JD, Maclean CJ, Vollmer WM, Johnson LR, Fong KO, Rodriguez BL, Masaki KH, Buist AS. Effects of smoking and smoking cessation on longitudinal decline in pulmonary function. Am J Respir Crit Care Med. 1995 Jun;151(6):1778-85. doi: 10.1164/ajrccm.151.6.7767520.
- [Background] Curb JD, Rodriguez BL, Burchfiel CM, Abbott RD, Chiu D, Yano K. Sudden death, impaired glucose tolerance, and diabetes in Japanese American men. Circulation. 1995 May 15;91(10):2591-5. doi: 10.1161/01.cir.91.10.2591. PMID 7743621
- [Background] Burchfiel CM, Sharp DS, Curb JD, Rodriguez BL, Hwang LJ, Marcus EB, Yano K. Physical activity and incidence of diabetes: the Honolulu Heart Program. Am J Epidemiol. 1995 Feb 15;141(4):360-8. doi: 10.1093/aje/141.4.360. PMID 7840114
- [Background] Petrovitch H, Curb JD, Bloom-Marcus E. Isolated systolic hypertension and risk of stroke in Japanese-American men. Stroke. 1995 Jan;26(1):25-9. doi: 10.1161/01.str.26.1.25. PMID 7839392
- [Background] Burchfiel CM, Curb JD, Rodriguez BL, Yano K, Hwang LJ, Fong KO, Marcus EB. Incidence and predictors of diabetes in Japanese-American men. The Honolulu Heart Program. Ann Epidemiol. 1995 Jan;5(1):33-43. doi: 10.1016/1047-2797(94)00038-u. PMID 7728283
- [Background] Abbott RD, Behrens GR, Sharp DS, Rodriguez BL, Burchfiel CM, Ross GW, Yano K, Curb JD. Body mass index and thromboembolic stroke in nonsmoking men in older middle age. The Honolulu Heart Program. Stroke. 1994 Dec;25(12):2370-6. doi: 10.1161/01.str.25.12.2370. PMID 7974575
- [Background] Rodriguez BL, Masaki K, Burchfiel C, Curb JD, Fong KO, Chyou PH, Marcus EB. Pulmonary function decline and 17-year total mortality: the Honolulu Heart Program. Am J Epidemiol. 1994 Sep 1;140(5):398-408. doi: 10.1093/oxfordjournals.aje.a117262. PMID 8067332
- [Background] Benfante R, Hwang LJ, Masaki K, Curb JD. To what extent do cardiovascular risk factor values measured in elderly men represent their midlife values measured 25 years earlier? A preliminary report and commentary from the Honolulu Heart Program. Am J Epidemiol. 1994 Aug 1;140(3):206-16. doi: 10.1093/oxfordjournals.aje.a117240. PMID 8030624
- [Background] Rodriguez BL, Curb JD, Burchfiel CM, Abbott RD, Petrovitch H, Masaki K, Chiu D. Physical activity and 23-year incidence of coronary heart disease morbidity and mortality among middle-aged men. The Honolulu Heart Program. Circulation. 1994 Jun;89(6):2540-4. doi: 10.1161/01.cir.89.6.2540. PMID 8205662
- [Background] Abbott RD, Rodriguez BL, Burchfiel CM, Curb JD. Physical activity in older middle-aged men and reduced risk of stroke: the Honolulu Heart Program. Am J Epidemiol. 1994 May 1;139(9):881-93. doi: 10.1093/oxfordjournals.aje.a117094. PMID 8166138
- [Background] Burchfiel CM, Curb JD, Rodriguez BL, Abbott RD, Chiu D, Yano K. Glucose intolerance and 22-year stroke incidence. The Honolulu Heart Program. Stroke. 1994 May;25(5):951-7. doi: 10.1161/01.str.25.5.951. PMID 8165689
- [Background] Benfante R, Yano K, Hwang LJ, Curb JD, Kagan A, Ross W. Elevated serum cholesterol is a risk factor for both coronary heart disease and thromboembolic stroke in Hawaiian Japanese men. Implications of shared risk. Stroke. 1994 Apr;25(4):814-20. doi: 10.1161/01.str.25.4.814. PMID 8160226
- [Background] Laws A, Marcus EB, Grove JS, Curb JD. Lipids and lipoproteins as risk factors for coronary heart disease in men with abnormal glucose tolerance: the Honolulu Heart Program. J Intern Med. 1993 Nov;234(5):471-8. doi: 10.1111/j.1365-2796.1993.tb00780.x. PMID 8228791
- [Background] Scherr PA, LaCroix AZ, Wallace RB, Berkman L, Curb JD, Cornoni-Huntley J, Evans DA, Hennekens CH. Light to moderate alcohol consumption and mortality in the elderly. J Am Geriatr Soc. 1992 Jul;40(7):651-7. doi: 10.1111/j.1532-5415.1992.tb01954.x. PMID 1607579
- [Background] Taylor JO, Cornoni-Huntley J, Curb JD, Manton KG, Ostfeld AM, Scherr P, Wallace RB. Blood pressure and mortality risk in the elderly. Am J Epidemiol. 1991 Sep 1;134(5):489-501. doi: 10.1093/oxfordjournals.aje.a116121. PMID 1897505
- [Background] Curb JD, Marcus EB. Body fat and obesity in Japanese Americans. Am J Clin Nutr. 1991 Jun;53(6 Suppl):1552S-1555S. doi: 10.1093/ajcn/53.6.1552S. PMID 2031486
- [Background] Foley DJ, Monjan AA, Masaki KH, Enright PL, Quan SF, White LR. Associations of symptoms of sleep apnea with cardiovascular disease, cognitive impairment, and mortality among older Japanese-American men. J Am Geriatr Soc. 1999 May;47(5):524-8. doi: 10.1111/j.1532-5415.1999.tb02564.x. PMID 10323643
- [Background] Galanis DJ, Harris T, Sharp DS, Petrovitch H. Relative weight, weight change, and risk of coronary heart disease in the Honolulu Heart Program. Am J Epidemiol. 1998 Feb 15;147(4):379-86. doi: 10.1093/oxfordjournals.aje.a009460. PMID 9508105
- [Background] Sharp DS, Masaki K, Burchfiel CM, Yano K, Schatz IJ. Prolonged QTc interval, impaired pulmonary function, and a very lean body mass jointly predict all-cause mortality in elderly men. Ann Epidemiol. 1998 Feb;8(2):99-106. doi: 10.1016/s1047-2797(97)00121-x. PMID 9491934
- [Background] Grove JS, Reed DM, Yano K, Hwang LJ. Variability in systolic blood pressure--a risk factor for coronary heart disease? Am J Epidemiol. 1997 May 1;145(9):771-6. doi: 10.1093/oxfordjournals.aje.a009169. PMID 9143206
- [Background] Burchfiel CM, Tracy RE, Chyou PH, Strong JP. Cardiovascular risk factors and hyalinization of renal arterioles at autopsy. The Honolulu Heart Program. Arterioscler Thromb Vasc Biol. 1997 Apr;17(4):760-8. doi: 10.1161/01.atv.17.4.760. PMID 9108792
- [Background] Burchfiel CM, Reed DM, Strong JP, Sharp DS, Chyou PH, Rodriguez BL. Predictors of myocardial lesions in men with minimal coronary atherosclerosis at autopsy. The Honolulu heart program. Ann Epidemiol. 1996 Mar;6(2):137-46. doi: 10.1016/1047-2797(95)00125-5. PMID 8775594
- [Background] Iribarren C, Sharp D, Burchfiel CM, Sun P, Dwyer JH. Association of serum total cholesterol with coronary disease and all-cause mortality: multivariate correction for bias due to measurement error. Am J Epidemiol. 1996 Mar 1;143(5):463-71. doi: 10.1093/oxfordjournals.aje.a008766. PMID 8610661
- [Background] Iribarren C, Reed DM, Chen R, Yano K, Dwyer JH. Low serum cholesterol and mortality. Which is the cause and which is the effect? Circulation. 1995 Nov 1;92(9):2396-403. doi: 10.1161/01.cir.92.9.2396. PMID 7586337
- [Background] Iribarren C, Sharp DS, Burchfiel CM, Petrovitch H. Association of weight loss and weight fluctuation with mortality among Japanese American men. N Engl J Med. 1995 Sep 14;333(11):686-92. doi: 10.1056/NEJM199509143331102. PMID 7637745
- [Background] Iribarren C, Reed DM, Wergowske G, Burchfiel CM, Dwyer JH. Serum cholesterol level and mortality due to suicide and trauma in the Honolulu Heart Program. Arch Intern Med. 1995 Apr 10;155(7):695-700. PMID 7695457
- [Background] Goldberg RJ, Burchfiel CM, Benfante R, Chiu D, Reed DM, Yano K. Lifestyle and biologic factors associated with atherosclerotic disease in middle-aged men. 20-year findings from the Honolulu Heart Program. Arch Intern Med. 1995 Apr 10;155(7):686-94. PMID 7695456
- [Background] Sharp DS, Rodriguez BL, Shahar E, Hwang LJ, Burchfiel CM. Fish consumption may limit the damage of smoking on the lung. Am J Respir Crit Care Med. 1994 Oct;150(4):983-7. doi: 10.1164/ajrccm.150.4.7921474.
- [Background] Kagan A, Popper J, Reed DM, MacLean CJ, Grove JS. Trends in stroke incidence and mortality in Hawaiian Japanese men. Stroke. 1994 Jun;25(6):1170-5. doi: 10.1161/01.str.25.6.1170. PMID 8202975
- [Background] Goldberg RJ, Burchfiel CM, Reed DM, Wergowske G, Chiu D. A prospective study of the health effects of alcohol consumption in middle-aged and elderly men. The Honolulu Heart Program. Circulation. 1994 Feb;89(2):651-9. doi: 10.1161/01.cir.89.2.651. PMID 8313554
- [Background] Yano K, Popper JS, Kagan A, Chyou PH, Grove JS. Epidemiology of stroke among Japanese men in Hawaii during 24 years of follow-up: the Honolulu Heart Program. Health Rep. 1994;6(1):28-38. English, French. PMID 7919086
- [Background] Yano K, Grove JS, Reed DM, Chun HM. Determinants of the prognosis after a first myocardial infarction in a migrant Japanese population. The Honolulu Heart Program. Circulation. 1993 Dec;88(6):2582-95. doi: 10.1161/01.cir.88.6.2582. PMID 8252669
- [Background] Burchfiel CM, Reed DM, Marcus EB, Strong JP, Hayashi T. Association of diabetes mellitus with coronary atherosclerosis and myocardial lesions. An autopsy study from the Honolulu Heart Program. Am J Epidemiol. 1993 Jun 15;137(12):1328-40. doi: 10.1093/oxfordjournals.aje.a116642. PMID 8333414
- [Background] Miller FD, Reed DM, MacLean CJ. Mortality and morbidity among blue and white collar workers in the Honolulu Heart Program cohort. Int J Epidemiol. 1993 Oct;22(5):834-7. doi: 10.1093/ije/22.5.834. PMID 8282462
- [Background] Benfante R. Studies of cardiovascular disease and cause-specific mortality trends in Japanese-American men living in Hawaii and risk factor comparisons with other Japanese populations in the Pacific region: a review. Hum Biol. 1992 Dec;64(6):791-805. PMID 1427739
- [Background] Frank JW, Reed DM, Grove JS, Benfante R. Will lowering population levels of serum cholesterol affect total mortality? Expectations from the Honolulu Heart Program. J Clin Epidemiol. 1992 Apr;45(4):333-46. doi: 10.1016/0895-4356(92)90034-k. PMID 1569429
- [Background] Reed D, Benfante R. Lipid and lipoprotein predictors of coronary heart disease in elderly men in the Honolulu Heart Program. Ann Epidemiol. 1992 Jan-Mar;2(1-2):29-34. doi: 10.1016/1047-2797(92)90034-n. PMID 1342261
- [Background] Reed D, Yano K. Predictors of arteriographically defined coronary stenosis in the Honolulu Heart Program. Comparisons of cohort and arteriography series analyses. Am J Epidemiol. 1991 Jul 15;134(2):111-22. doi: 10.1093/oxfordjournals.aje.a116063. PMID 1862795
- [Background] Benfante R, Reed D, Frank J. Does cigarette smoking have an independent effect on coronary heart disease incidence in the elderly? Am J Public Health. 1991 Jul;81(7):897-9. doi: 10.2105/ajph.81.7.897. PMID 2053668
- [Background] Stemmermann GN, Chyou PH, Kagan A, Nomura AM, Yano K. Serum cholesterol and mortality among Japanese-American men. The Honolulu (Hawaii) Heart Program. Arch Intern Med. 1991 May;151(5):969-72. PMID 2025146
- [Background] Reed D, Marcus E, Hayashi T. Smoking as a predictor of atherosclerosis in the Honolulu Heart Program. Adv Exp Med Biol. 1990;273:17-25. doi: 10.1007/978-1-4684-5829-9_3. No abstract available. PMID 2288273
- [Background] Petrovitch H, White L, Masaki KH, Ross GW, Abbott RD, Rodriguez BL, Lu G, Burchfiel CM, Blanchette PL, Curb JD. Influence of myocardial infarction, coronary artery bypass surgery, and stroke on cognitive impairment in late life. Am J Cardiol. 1998 Apr 15;81(8):1017-21. doi: 10.1016/s0002-9149(98)00082-4. PMID 9576163
- [Background] Abbott RD, Petrovitch H, Rodriguez BL, Yano K, Schatz IJ, Popper JS, Masaki KH, Ross GW, Curb JD. Ankle/brachial blood pressure in men >70 years of age and the risk of coronary heart disease. Am J Cardiol. 2000 Aug 1;86(3):280-4. doi: 10.1016/s0002-9149(00)00914-0. PMID 10922433
- [Background] Kalmijn S, Foley D, White L, Burchfiel CM, Curb JD, Petrovitch H, Ross GW, Havlik RJ, Launer LJ. Metabolic cardiovascular syndrome and risk of dementia in Japanese-American elderly men. The Honolulu-Asia aging study. Arterioscler Thromb Vasc Biol. 2000 Oct;20(10):2255-60. doi: 10.1161/01.atv.20.10.2255. PMID 11031212
- [Background] Kardaun JW, White L, Resnick HE, Petrovitch H, Marcovina SM, Saunders AM, Foley DJ, Havlik RJ. Genotypes and phenotypes for apolipoprotein E and Alzheimer disease in the Honolulu-Asia aging study. Clin Chem. 2000 Oct;46(10):1548-54. PMID 11017931
- [Background] Foley DJ, Masaki KH, Ross GW, White LR. Driving cessation in older men with incident dementia. J Am Geriatr Soc. 2000 Aug;48(8):928-30. doi: 10.1111/j.1532-5415.2000.tb06889.x. PMID 10968296
- [Background] Petrovitch H, White LR, Izmirilian G, Ross GW, Havlik RJ, Markesbery W, Nelson J, Davis DG, Hardman J, Foley DJ, Launer LJ. Midlife blood pressure and neuritic plaques, neurofibrillary tangles, and brain weight at death: the HAAS. Honolulu-Asia aging Study. Neurobiol Aging. 2000 Jan-Feb;21(1):57-62. doi: 10.1016/s0197-4580(00)00106-8. PMID 10794849
- [Background] Ceria CD, Masaki KH, Rodriguez BL, Chen R, Yano K, Curb JD. The relationship of psychosocial factors to total mortality among older Japanese-American men: the Honolulu Heart Program. J Am Geriatr Soc. 2001 Jun;49(6):725-31. doi: 10.1046/j.1532-5415.2001.49148.x. PMID 11454110
- [Background] Yano K, Grove JS, Chen R, Rodriguez BL, Curb JD, Tracy RP. Plasma fibrinogen as a predictor of total and cause-specific mortality in elderly Japanese-American men. Arterioscler Thromb Vasc Biol. 2001 Jun;21(6):1065-70. doi: 10.1161/01.atv.21.6.1065. PMID 11397721
- [Background] Sharp DS, Burchfiel CM, Rodriguez BL, Sharrett AR, Sorlie PD, Marcovina SM. Apolipoprotein A-1 predicts coronary heart disease only at low concentrations of high-density lipoprotein cholesterol: an epidemiological study of Japanese-Americans. Int J Clin Lab Res. 2000;30(1):39-48. doi: 10.1007/s005990070032. PMID 10984131
- [Background] Abbott RD, Curb JD, Rodriguez BL, Masaki KH, Yano K, Schatz IJ, Ross GW, Petrovitch H. Age-related changes in risk factor effects on the incidence of coronary heart disease. Ann Epidemiol. 2002 Apr;12(3):173-81. doi: 10.1016/s1047-2797(01)00309-x. PMID 11897175
- [Background] Rodriguez BL, D'Agostino R, Abbott RD, Kagan A, Burchfiel CM, Yano K, Ross GW, Silbershatz H, Higgins MW, Popper J, Wolf PA, Curb JD. Risk of hospitalized stroke in men enrolled in the Honolulu Heart Program and the Framingham Study: A comparison of incidence and risk factor effects. Stroke. 2002 Jan;33(1):230-6. doi: 10.1161/hs0102.101081. PMID 11779915
- [Background] Abbott RD, Rodriguez BL, Petrovitch H, Yano K, Schatz IJ, Popper JS, Masaki KH, Ross GW, Curb JD. Ankle-brachial blood pressure in elderly men and the risk of stroke: the Honolulu Heart Program. J Clin Epidemiol. 2001 Oct;54(10):973-8. doi: 10.1016/s0895-4356(01)00373-0. PMID 11576807
- [Background] Rodriguez BL, Abbott RD, Fujimoto W, Waitzfelder B, Chen R, Masaki K, Schatz I, Petrovitch H, Ross W, Yano K, Blanchette PL, Curb JD; American Diabetes Association; World Health Organization. The American Diabetes Association and World Health Organization classifications for diabetes: their impact on diabetes prevalence and total and cardiovascular disease mortality in elderly Japanese-American men. Diabetes Care. 2002 Jun;25(6):951-5. doi: 10.2337/diacare.25.6.951. PMID 12032097
- [Background] Laurin D, Foley DJ, Masaki KH, White LR, Launer LJ. Vitamin E and C supplements and risk of dementia. JAMA. 2002 Nov 13;288(18):2266-8. doi: 10.1001/jama.288.18.2266. No abstract available. PMID 12425703
- [Background] Curb JD, Abbott RD, Rodriguez BL, Sakkinen P, Popper JS, Yano K, Tracy RP. C-reactive protein and the future risk of thromboembolic stroke in healthy men. Circulation. 2003 Apr 22;107(15):2016-20. doi: 10.1161/01.CIR.0000065228.20100.F7. Epub 2003 Apr 7. PMID 12681999
- [Background] Abbott RD, Ando F, Masaki KH, Tung KH, Rodriguez BL, Petrovitch H, Yano K, Curb JD. Dietary magnesium intake and the future risk of coronary heart disease (the Honolulu Heart Program). Am J Cardiol. 2003 Sep 15;92(6):665-9. doi: 10.1016/s0002-9149(03)00819-1. PMID 12972103
- [Background] Petrovitch H, Ross GW, Abbott RD, Sanderson WT, Sharp DS, Tanner CM, Masaki KH, Blanchette PL, Popper JS, Foley D, Launer L, White LR. Plantation work and risk of Parkinson disease in a population-based longitudinal study. Arch Neurol. 2002 Nov;59(11):1787-92. doi: 10.1001/archneur.59.11.1787. PMID 12433267
- [Background] Abbott RD, Curb JD, Rodriguez BL, Masaki KH, Popper JS, Ross GW, Petrovitch H. Age-related changes in risk factor effects on the incidence of thromboembolic and hemorrhagic stroke. J Clin Epidemiol. 2003 May;56(5):479-86. doi: 10.1016/s0895-4356(02)00611-x. PMID 12812823
- [Background] Curb JD, Abbott RD, Rodriguez BL, Masaki KH, Chen R, Popper JS, Petrovitch H, Ross GW, Schatz IJ, Belleau GC, Yano K. High density lipoprotein cholesterol and the risk of stroke in elderly men: the Honolulu heart program. Am J Epidemiol. 2004 Jul 15;160(2):150-7. doi: 10.1093/aje/kwh177. PMID 15234936
- [Background] Curb JD, Abbott RD, Rodriguez BL, Masaki K, Chen R, Sharp DS, Tall AR. A prospective study of HDL-C and cholesteryl ester transfer protein gene mutations and the risk of coronary heart disease in the elderly. J Lipid Res. 2004 May;45(5):948-53. doi: 10.1194/jlr.M300520-JLR200. Epub 2004 Feb 16. PMID 14967821
- [Background] Abbott RD, White LR, Ross GW, Masaki KH, Curb JD, Petrovitch H. Walking and dementia in physically capable elderly men. JAMA. 2004 Sep 22;292(12):1447-53. doi: 10.1001/jama.292.12.1447. PMID 15383515
- [Background] Yano K, Reed DM, MacLean CJ. Serum cholesterol and hemorrhagic stroke in the Honolulu Heart Program. Stroke. 1989 Nov;20(11):1460-5. doi: 10.1161/01.str.20.11.1460. PMID 2815179
- [Background] Yano K, MacLean CJ. The incidence and prognosis of unrecognized myocardial infarction in the Honolulu, Hawaii, Heart Program. Arch Intern Med. 1989 Jul;149(7):1528-32. PMID 2742427
- Available data/document: Individual Participant Data Set: HHP — http://biolincc.nhlbi.nih.gov/studies/hhp/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Data Coding Manuals — http://biolincc.nhlbi.nih.gov/studies/hhp/